CLINICAL TRIAL: NCT05267392
Title: Neoadjuvant Immunotherapy With Durvalumab (MEDI4736) in Non-Surgical Early Stage or Locally Advanced Non-Small Cell Lung Cancer (NSCLC) Followed by Radical Radiotherapy or Chemoradiotherapy
Acronym: IDEAR
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Instituto Portugues de Oncologia, Francisco Gentil, Porto (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ESR-18-13828; 2019-002884-90 (EudraCT Number)
Record Dates: First submitted 2021-12-13; First posted 2022-03-04 (Actual); Last update posted 2022-03-04 (Actual); Status verified 2021-12

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Non-Small Cell Lung Cancer (NSCLC); PD1/PD-L1; anti-PD1/PD-L1 blockade; Non-Surgical Early Stage or Locally Advanced NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — durvalumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Durvalumab (Experimental): All subjects enrolled in the study will receive open-label neoadjuvant durvalumab 1500 mg followed by standard of care RT/RCT
  Interventions: Drug: Durvalumab; Other: standard of care RT/RCT

INTERVENTIONS:
Drug: Durvalumab — Patients will receive 1500 mg of durvalumab (MEDI4736) via IV infusion
Other: standard of care RT/RCT — standard of care RT/RCT

SUMMARY:
This study proposes to evaluate the safety and efficacy of an anti-PD-L1 (durvalumab) agent as neoadjuvant therapy in patients diagnosed with localized NSCLC who are planned to undergo radical RT or CRT. The hypothesis to be tested for the primary objective is that the treatment of durvalumab followed by RT/CRT will be safe and well tolerated in subjects with NSCLC.

DETAILED DESCRIPTION:
Targeting the PD1/PD-L1 pathway has demonstrated activity in patients with several advanced malignancies. Treatment with anti-PD1/PD-L1 blockade in advanced and, more recently, locally advanced NSCLC, is already standard of care. The positive outcomes of durvalumab following CRT emphasized the potential of immunotherapy integration in multimodality treatment strategies and in earlier phases of the disease, leading to the first immune checkpoint inhibitor approval in non-metastatic setting in NSCLC. Furthermore, growing evidence is pointing to the efficacy of neoadjuvant treatments in NSCLC. This study proposes to evaluate the safety and efficacy of an anti-PD-L1 (durvalumab) agent as neoadjuvant therapy in patients diagnosed with localized NSCLC who are planned to undergo radical RT or CRT.

The hypothesis to be tested for:

* Primary objective: To evaluate the safety, as assessed by incidence of dose limiting toxicity (DLT), of durvalumab followed by RT/CRT in patients with early stage or locally advanced, unresectable NSCLC who are planned to undergo radical RT or CRT.
* Secondary Objectives: To evaluate the safety, the efficacy and the feasibility of durvalumab followed by RT/CRT.
* Exploratory Objectives: To assess the Quality of Life (QoL) using SF-36v2 and EQ-5D-5L and to assess blood and tumor tissue for potential biomarkers which predict and/or correlate with clinical outcomes.

ELIGIBILITY:
Inclusion Criteria

1. Patients capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in the protocol.
2. Age ≥ 18 years at time of screening.
3. ECOG performance status of 0 or 1.
4. Life expectancy of at least 12 weeks.
5. Body weight >30 kg.
6. Histologically documented NSCLC.
7. Clinical Stage IIIA NSCLC eligible for RT (Initial work-up including PET-CT and brain MRI or brain CT for staging); patients with stage IB (≥ 4 cm)-IIIA NSCLC that are not considered for surgical treatment by the clinical team (e.g.: due to comorbidities) or by patient choice, but are eligible for radical RT or CRT can be proposed for inclusion.
8. Measurable disease, as defined by RECIST.
9. Adequate normal organ and marrow function defined by the following laboratory results obtained within 14 days prior to durvalumab administration:

   1. Hemoglobin ≥ 9.0 g/dL.
   2. White blood cell (WBC) counts > 2.5 x 109/L.
   3. Absolut neutrophil count (ANC) ≥ 1.5 x 109/L (without granulocyte colony-stimulating factor support within 2 weeks prior to durvalumab treatment).
   4. Lymphocyte count ≥ 0.5 x 109/L.
   5. Platelet count ≥100 x 109/L.
   6. AST, ALT, and alkaline phosphatase ≤ 2.5 x the institutional upper limit of normal (ULN).
   7. Serum bilirubin ≤ 1.5 x ULN. Patients with known Gilbert disease who have serum bilirubin level ≤ 3 x ULN may be enrolled.
   8. International Normalized Ratio (INR) and activated Partial Thromboplastin Time (aPTT) ≤ 1.5 x ULN -This applies only to patients who are not receiving therapeutic anticoagulation; patients receiving therapeutic anticoagulation should be on a stable dose.
   9. Serum albumin ≥2.5 g/dL.
   10. Calcemia ≤2.65 mmol/L or Ca ≤10 mg/dL.
   11. Measured creatinine clearance (CL) >40 mL/min or Calculated creatinine CL>40 mL/min by the Cockcroft-Gault formula (Cockcroft and Gault 1976) or by 24-hour urine collection for determination of creatinine clearance.
10. Patient is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up.
11. Evidence of post-menopausal status or negative urinary or serum pregnancy test for female pre-menopausal patients. Women will be considered post-menopausal if they have been amenorrhoeic for 12 months without an alternative medical cause. The following age-specific requirements apply:

    1. Women <50 years of age would be considered post-menopausal if they have been amenorrhoeic for 12 months or more following cessation of exogenous hormonal treatments and if they have luteinizing hormone and follicle-stimulating hormone levels in the post-menopausal range for the institution or underwent surgical sterilization (bilateral oophorectomy or hysterectomy).
    2. Women ≥50 years of age would be considered post-menopausal if they have been amenorrhoeic for 12 months or more following cessation of all exogenous hormonal treatments, had radiation-induced menopause with last menses >1 year ago, had chemotherapy-induced menopause with last menses >1 year ago, or underwent surgical sterilization (bilateral oophorectomy, bilateral salpingectomy or hysterectomy).
12. Women of Childbearing Potential must be willing to use 1 highly effective method of contraception, or to abstain from sexual activity, from the time of screening throughout the total duration of the drug treatment and for 3 months after the last session of RT/CRT. Non-sterilized male partners of a female patient of childbearing potential must use male condom plus spermicide throughout this period.
13. Non-sterilized male patients who are not abstinent and intend to be sexually active with a female partner of childbearing potential must use a male condom plus spermicide from the time of screening throughout the total duration of the drug treatment and for 3 months after the last session of RT/CRT. Male patients should refrain from sperm donation throughout this period. Female partners (of childbearing potential) of male patients must also use a highly effective method of contraception throughout this period.

    ------

Exclusion Criteria

1. Participation in another clinical study with an investigational product during the last 4 weeks prior to durvalumab administration.
2. Concurrent enrolment in another clinical study, unless it is an observational (non-interventional) clinical study or during the follow-up period of an interventional study.
3. Any unresolved toxicity NCI CTCAE, Version 5, Grade ≥2 from previous anticancer therapy with the exception of alopecia, vitiligo, and the laboratory values defined in the inclusion criteria:

   1. Patients with Grade ≥2 neuropathy will be evaluated on a case-by-case basis after consultation with the Study Physician.
   2. Patients with irreversible toxicity not reasonably expected to be exacerbated by treatment with durvalumab may be included only after consultation with the Study Physician.
4. Any concurrent chemotherapy, investigational product, biologic, or hormonal therapy for cancer treatment. Concurrent use of hormonal therapy for non-cancer-related conditions (e.g., hormone replacement therapy) is acceptable.
5. Prior chemotherapy or radiation therapy for lung cancer.
6. Major surgical procedure (as defined by the Investigator) within 28 days prior to the first dose of investigational product.
7. History of allogenic organ transplantation.
8. Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [e.g., colitis or Crohn's disease], diverticulitis [with the exception of diverticulosis], systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc.]). The following are exceptions to this criterion:

   1. Patients with vitiligo or alopecia.
   2. Patients with hypothyroidism (e.g., following Hashimoto syndrome) stable on hormone replacement.
   3. Any chronic skin condition that does not require systemic therapy.
   4. Patients without active disease in the last 5 years.
   5. Patients with celiac disease controlled by diet alone.
9. Uncontrolled intercurrent illness, including but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, interstitial lung disease, serious chronic gastrointestinal conditions associated with diarrhea, or psychiatric illness/social situations that would limit compliance with study requirement, substantially increase risk of incurring AEs or compromise the ability of the patient to give written informed consent.
10. History of another primary malignancy except for:

    1. Malignancy treated with curative intent and with no known active disease ≥5 years before the first dose of investigational product and of low potential risk for recurrence.
    2. Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease
    3. Adequately treated carcinoma in situ without evidence of disease.
11. History of leptomeningeal carcinomatosis.
12. History of active primary immunodeficiency.
13. Active infection including tuberculosis (clinical evaluation that includes clinical history, physical examination and radiographic findings, and TB testing in line with local practice), hepatitis B (known positive HBV surface antigen (HBsAg) result), hepatitis C, or human immunodeficiency virus (positive HIV 1/2 antibodies). Patients with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody [anti-HBc] and absence of HBsAg) are eligible. Patients positive for hepatitis C (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV RNA.
14. Current or prior use of immunosuppressive medication within 14 days before the administration of durvalumab. The following are exceptions to this criterion:

    1. Intranasal, inhaled, topical steroids, or local steroid injections (e.g., intra articular injection).
    2. Systemic corticosteroids at physiologic doses not to exceed 10 mg/day of prednisone or its equivalent.
    3. Steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication).
15. Receipt of live attenuated vaccine within 30 days prior to durvalumab infusion. Note: Patients, if enrolled, should not receive live vaccine up to 30 days after durvalumab infusion.
16. Female patients who are pregnant or breastfeeding or male or female patients of reproductive potential who are not willing to employ effective birth control from screening to 3 months after the last session of RT/CRT.
17. Known allergy or hypersensitivity to any of the study drugs or any of its excipients.
18. Prior randomization or treatment in a previous durvalumab clinical study regardless of treatment arm assignment.
19. History of severe allergic, anaphylactic, or other hypersensitivity reactions to chimeric or humanized antibodies.
20. History of idiopathic pulmonary fibrosis, organizing pneumonia (e.g., bronchiolitis obliterans), drug-induced pneumonitis, idiopathic pneumonitis, or evidence of active pneumonitis on screening chest CT scan.
21. Severe infections within 4 weeks prior to screening, including but not limited to hospitalization for complications of infection, bacteremia, or severe pneumonia.
22. Signs or symptoms of infection within 2 weeks prior to screening.
23. History of any hematological disease not considered in complete remission for at least 5 years before screening.
24. Any other diseases, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that may affect the interpretation of the results or render the patient at high risk from treatment complications.
25. Judgment by the investigator that the patient is unsuitable to participate in the study and the patient is unlikely to comply with study procedures, restrictions and requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-02-16 (Actual); Primary Completion 2023-07 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of Dose-Limiting Toxicity (DLT) | Through study development up to 5 - 6 weeks after the last session of RT/CRT for each enrolled patient
  Rate of patients without Dose-Limiting Toxicity (DLT) evaluated from durvalumab administration until 5 - 6 weeks after the last session of RT/CRT.

SECONDARY OUTCOMES:
Safety of durvalumab followed by RT/CRT | Through study development up to 17 weeks for each enrolled patient
  Presence of adverse events (AEs) assessed by (CTCAE) version 5.0
objective response rate | Through study development up to 17 weeks for each enrolled patient
  percentage of patients having a complete response or a partial response as measured by RECIST 1.1.
Pathologic response rate | Through study development up to 17 weeks for each enrolled patient
  Patients in whom tumor "downstaging" was achieved and making the patient eligible for surgery.
feasibility of durvalumab followed by RT/CRT | Through study development up to 3 years
  proportion of enrolled patients starting RT/CRT within 4 - 5 weeks after durvalumab administration and proportion of enrolled patients completing the clinical trial.

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto Português de Oncologia do Porto FG, EPE (IPO-Porto), Porto, Portugal